CLINICAL TRIAL: NCT01509079
Title: Phase 2 Study Vitamin D3 Effects on Musculoskeletal Symptoms With Use of Aromatase Inhibitors
Brief Title: Vitamin D3 Effects on Musculoskeletal Symptoms With Use of Aromatase Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: University of Minnesota (Other); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 03962-10C
Record Dates: First submitted 2011-12-12; First posted 2012-01-12 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2015-10

CONDITIONS: Muscle Pain; Joint Pain
MeSH Terms: conditions — Myalgia; Arthralgia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 4000 IU (Experimental)
  Interventions: Drug: Vitamin D3
- Vitamin D3 600 IU (Active Comparator)
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Cholecalciferol capsule, 4000IU, daily for 6 months
  Arms: Vitamin D3 4000 IU
Drug: Vitamin D3 — cholecalciferol capsule, 600 IU, daily for 6 months
  Arms: Vitamin D3 600 IU

SUMMARY:
The Purpose of this study is to determine whether vitamin D3 supplements will decrease the muscle and bone pain that are reported by women who take Aromatase Inhibitors.

DETAILED DESCRIPTION:
This project will determine the efficacy of vitamin D3 supplements for reducing side effects of treatment with aromatase inhibitors in women with a history of breast cancer that have no evidence of current disease. The aromatase inhibitors (AI) have become a critical component of adjuvant therapy for this population, but they cause bone pain, joint pain, joint stiffness, and muscle weakness in approximately 40% of patients. These symptoms, referred to as aromatase inhibitor-associated musculoskeletal symptoms (AIMSS), decrease quality of life and medication adherence. Identifying effective ways to decrease these symptoms may allow for longer and more adherent medication use and thus may improve disease-free survival. We hypothesize that vitamin D3 may decrease symptoms associated with the use of aromatase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Women with a history of stage I-IIIa invasive breast cancer
* History of hormone-receptor positive cancer (either ER + or PR + or both)
* Are prescribed and are taking anastrozole, letrozole or exemestane for at least one month and have at least 7 months of AI treatment remaining
* Are experiencing AIMSS

Exclusion Criteria:

* Unable to read or understand English
* History of psychiatric disability affecting informed consent or compliance with drug intake
* Malabsorption syndrome or inability to take oral medication
* Has less than 7 months of AI therapy remaining

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice C. Shapiro, PhD RD, Principal Investigator — Park Nicollet Health Services
Locations (1):
- Park Nicollet Frauenshuh Cancer Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Shapiro AC, Adlis SA, Robien K, Kirstein MN, Liang S, Richter SA, Lerner RE. Randomized, blinded trial of vitamin D3 for treating aromatase inhibitor-associated musculoskeletal symptoms (AIMSS). Breast Cancer Res Treat. 2016 Feb;155(3):501-12. doi: 10.1007/s10549-016-3710-6. Epub 2016 Feb 11. PMID 26868123

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D3 4000 IU | Vitamin D3 600 IU
Started | 57 | 59
Completed | 57 | 56
Not Completed | 0 | 3
Not completed — Lack of Efficacy | 0 | 2
Not completed — started an excluded medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 4000 IU | Vitamin D3 600 IU | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8.4) | 60.3 (9.3) | 60.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 113
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 57 | 56 | 113

OUTCOME MEASURES:

1. Primary Outcome: Change in Musculoskeletal Symptom Sub-scale on the Breast Cancer Prevention Trial Symptom Scale
Description: The MS subscale is a self-reported measure on a scale of 0 to 4, with lower score indicating less arthralgia/myalgia
Time Frame: baseline to 6 months
Population: Only participants who provided data at both time points are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vitamin D3 4000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 57 | 55
units on a scale | -0.2 (0.7) | -0.5 (0.9)
Statistical Analysis 1: Comparison: Vitamin D3 4000 IU vs Vitamin D3 600 IU; Test type: Superiority or Other; p = 0.38, ANOVA

2. Primary Outcome: Change in Hand Grip Strength
Time Frame: baseline to 6 months
Population: only data from participants that were collected at both time points is included
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Vitamin D3 4000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 54 | 53
pounds | 1.8 (10.6) | 1.0 (7.6)

3. Secondary Outcome: Change in PROMIS Physical Functioning Questionnaire
Description: PROMIS measures physical functioning on the short form and higher scores reflect better physical functioning with 10 questions on daily activities of life on a Likert scale ranging from 5 (no problem performing activity) to 1 (cannot do activity). Range on this measure is from 50 (best)-10 (worst).
Time Frame: baseline to 6 months
Population: only data from participants with measures at both time points are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vitamin D3 4000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 57 | 55
units on a scale | 0.6 (4.9) | 1.7 (6.9)

4. Secondary Outcome: Average Percent Adherence to Vitamin D Interventio
Description: adherence measured with pill counts for the vitamin D at predesignated study timepoints: baseline (after run-in), 3 months and 6 months
Time Frame: average for all study ppts for: screening to baseline; baseline to 3 months; 3 month to 6 months
Measure: Number; unit: % of adherence for each treatment arm
Arm/Group | Vitamin D3 4000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 57 | 56
% of adherence for each treatment arm | 95 | 95

5. Secondary Outcome: Serum Estradiol Concentrations
Time Frame: baseline and 6 months
Population: only participants whose serum was obtained at both time points are included
Measure: Geometric Mean (Standard Error); unit: pg/ml
Arm/Group | Vitamin D3 4000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 52 | 50
pg/ml
  Baseline | 2.83 (0.1) | 2.77 (0.1)
  6 months | 2.94 (0.16) | 3.0 (0.12)

6. Secondary Outcome: Change in Steady State Concentrations of Serum Anastrazole and Letrozole
Description: Difference in steady state concentrations in plasma from baseline to 6 months
Time Frame: baseline to 6 months
Population: Only study participants with baseline and 6 month blood samples available were analyzed
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Vitamin D3 4000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 47 | 48
mg/L
  anastrozole | -1.31 (10.67) | 2.4 (5.36)
  letrozole | 2.16 (9.69) | -0.83 (16.4)

7. Secondary Outcome: Whole Body Bone Mineral Density
Description: GLM Mean and standard deviation of Whole Body Bone Mineral Density (grams/cm2) of Trial Participants by Treatment Arm after controlling for bisphosphonate use
Time Frame: From Baseline and 6 months of D3 supplementation
Measure: Geometric Least Squares Mean (Standard Deviation); unit: gm/cm2
Arm/Group | Vitamin D3 4000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 53 | 54
gm/cm2 | 1.1 (0.12) | 1.12 (0.13)

8. Secondary Outcome: Vitamin D Binding Protein Genotype
Time Frame: Baseline
Population: Due to funding limitations, this secondary aim was not collected and analyzed in these groups
Arm/Group | Vitamin D3 4000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were collected with regard to the organ system
Arm/Group | Vitamin D3 4000 IU | Vitamin D3 600 IU
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 35/57 | 32/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D3 4000 IU (N=57) | Vitamin D3 600 IU (N=56)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 10 | 10
Gastrointestinal complaints (Gastrointestinal disorders) | 12 | 7
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 5 | 3
Surgical and medical procedures (Surgical and medical procedures) | 4 | 1
Nervous system disorders (Nervous system disorders) | 7 | 3
Respiratory (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Skin problems (Skin and subcutaneous tissue disorders) | 5 | 5
Cardiac (Cardiac disorders) | 2 | 3
General (General disorders) | 3 | 1
Reproductive and breast issues (Reproductive system and breast disorders) | 2 | 5
Injuries (Injury, poisoning and procedural complications) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No